CLINICAL TRIAL: NCT01609348
Title: Venlafaxine for Depression in Alzheimer's Disease
Brief Title: Venlafaxine for Depression in Alzheimer's Disease (DIADs-3)
Acronym: DIADs-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00066043
Record Dates: First submitted 2012-04-27; First posted 2012-06-01 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease; Depression
Keywords: Depression; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venlafaxine (Active Comparator): 225 mg daily over 12 weeks
  Interventions: Drug: Venlafaxine
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Capsule matching active drug to be taken once a day for 12 weeks
  Arms: Sugar pill
Drug: Venlafaxine — 225 mg daily for 12 weeks
  Arms: Venlafaxine

SUMMARY:
This study will test the use of venlafaxine to treat the depression in Alzheimer's Disease. Venlafaxine works by increasing natural substances in the brain (serotonin and norepinephrine) that help maintain mental balance. Alzheimer's disease (AD) is the commonest neurodegenerative disease of aging and the cause of major financial and emotional burden to patients, families and caregivers, and society. Depression is a very common symptom of AD, affecting as many as 50% of patients over their illness. Depression in AD (Alzheimer's disease) contributes greatly to patient disability and caregiver distress. Neither psychosocial interventions nor psychotropic medications have proven effective to date for the treatment of depression in AD.Venlafaxine is approved by the U.S. Food and Drug Administration (FDA) for the treatment of major depression but it is not known whether or not it can help depression in Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Dementia due to Alzheimer's disease by Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-IV (TR) criteria (90), with a Mini-Mental State Exam (MMSE) (82) score of 10-26 inclusive;
* Depression as defined by the National Institute of Mental Health (NIMH) Consensus Criteria,
* Clinical Dementia Rating Scale of 1 "mild" or 2 "moderate". Ratings of 3 "severe" will be excluded because many of the instruments lack validity in the presence of severe cognitive impairment, particularly language deficits.
* Sufficiently good health to be treated using the study protocol in usual care circumstances;
* Patient or surrogate and caregiver provides informed consent for participation in the study;
* A caregiver is available who spends at least 10 hours per week with the patient, supervises her care, and is willing to accompany the patient to study visits and to provide information about the patient.
* Female participants must be at least 2 years post menopause or surgically sterilized. Exclusion Criteria
* Presence of a brain disease that might otherwise fully explain the presence of dementia, such as stroke, Parkinson's disease, traumatic brain injury, multiple sclerosis, and similar neurologic diseases;
* Clinically significant psychosis that requires antipsychotic treatment; -Treatment with venlafaxine is contraindicated in the opinion of the attending psychiatrist, for example if there is a prior history of dangerous or -unacceptable side effects when treated with venlafaxine;
* Failure of treatment with venlafaxine in the past for depression after convincing evidence of a "good trial," for example 8 weeks at the highest tolerated dose;
* Treatment for a condition or with a medication that would prohibit the safe concurrent use of venlafaxine (specifically including systolic blood pressure > 180 mm Hg or diastolic blood pressure > 100 mm Hg);
* Diagnosis of congenital long Q-T syndrome
* The patient requires psychiatric hospitalization for depression or is suicidal;
* Initiation, discontinuation or dose changes in cholinesterase inhibitor or memantine use within the 4 weeks prior to screening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins at Bayview, Baltimore, Maryland
  - Reading Hospital, West Reading, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venlafaxine | Sugar Pill
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine | Sugar Pill | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Dose Response Using the Modified Alzheimer's Disease (AD) Cooperative Study-Clinical Global Impression of Change.
Description: Treatment will be considered efficacious if the proportion of worse categories (including 'minimal worsening', 'moderate worsening', or 'marked worsening') is lower under treatment than control on the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change.
  Clinical Global Impression of Change: This is a 7-item score ranging from "markedly worse" to "markedly improved". It is assessed by the study clinician who interviews both participant and informant and makes an informed judgment how to incorporate their input
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Venlafaxine | Sugar Pill
Number analyzed (Participants) | 3 | 2
Participants
  Marked improvement according to CGI | 2 | 0
  Moderate improvement according to CGI | 1 | 2

ADVERSE EVENTS:
Arm/Group | Venlafaxine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine (N=3) | Sugar Pill (N=2)
Hypokalemia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine (N=3) | Sugar Pill (N=2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Low potassium (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes